CLINICAL TRIAL: NCT00001104
Title: A Placebo Controlled Trial To Evaluate Zidovudine (ZDV) in the Treatment of Human Immunodeficiency Virus (HIV) Infection in Hemophilic Patients
Brief Title: A Study of Zidovudine in HIV-Infected Patients Who Have Hemophilia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 036; 11012 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Sex Behavior; T-Lymphocytes; HIV Antibodies; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Hemophilia A
MeSH Terms: conditions — HIV Infections; Sexual Behavior; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Hemophilia A | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
Study A: To determine whether treatment with zidovudine (ZDV) will delay or change the disease process in hemophilic patients who have HIV infection with no symptoms. The major clinical question is whether patients who receive chronic ZDV therapy will have a delay in the development of AIDS or AIDS-related complex (ARC). The pharmacokinetics (blood levels) of ZDV in hemophilic patients will also be studied.

Study B: To determine if ZDV therapy changes the risk of a hemophiliac transmitting HIV to his wife or other female sexual partner. To determine the effectiveness of counseling and education on the behaviors of the wives that place them at risk for HIV infection. To determine if antibodies to HIV either appear or disappear from the blood of any of the wives during the study.

Study A: Individuals who are infected with HIV can benefit from therapy with an effective anti-AIDS virus agent. ZDV is a potent inhibitor of HIV in vitro (test tube) and is safe in humans at the dose planned. It may be effective in preventing the development of AIDS or ARC in hemophiliacs who have the HIV antibody in their blood. The pharmacokinetic studies are especially important because the high prevalence of hepatic disease in this population may affect the metabolism and blood levels of ZDV.

Study B: HIV is transmitted by sexual contact, and wives of infected hemophilic patients have become infected during long-term sexual relationships. Transmission of the virus does not occur during casual family contact. This study will aid in determining if therapy influences the transmission of HIV, because the wives of hemophiliacs generally have no risk for HIV infection other than sexual contact with their spouse.

DETAILED DESCRIPTION:
Study A: Individuals who are infected with HIV can benefit from therapy with an effective anti-AIDS virus agent. ZDV is a potent inhibitor of HIV in vitro (test tube) and is safe in humans at the dose planned. It may be effective in preventing the development of AIDS or ARC in hemophiliacs who have the HIV antibody in their blood. The pharmacokinetic studies are especially important because the high prevalence of hepatic disease in this population may affect the metabolism and blood levels of ZDV.

Study B: HIV is transmitted by sexual contact, and wives of infected hemophilic patients have become infected during long-term sexual relationships. Transmission of the virus does not occur during casual family contact. This study will aid in determining if therapy influences the transmission of HIV, because the wives of hemophiliacs generally have no risk for HIV infection other than sexual contact with their spouse.

Study A: Patients selected for the study are randomly assigned to placebo (inactive medication) or ZDV taken every 4 hours while the patient is awake for a total of 5 doses per day. The patient's immune function and clinical condition are monitored with periodic virus cultures, p24 antigen assays, estimates of lymphocyte type and numbers, cell surface markers, and frequent clinical evaluations to see if these are markers of drug efficacy. Patients continue on their regimen until the final analysis of the data, which could occur up to 3 years after the last patient is entered into the study. Amendment: Based on data from ACTG 019 this protocol has been closed to further accrual. All patients entered in this study will be unblinded as to treatment received. Patients will be informed of results of ACTG 019 and be requested to sign a modified statement of consent approved by the local Institutional Review Board. All patients currently receiving study therapy will be offered open-label ZDV. Patients temporarily discontinued from study therapy at this time will be offered open-label ZDV when toxicity resolves (less than or equal to Grade 2 hemoglobin or neutrophil toxicity, less than or equal to Grade 1 all other toxicities). Patients who have been permanently discontinued from study therapy will not be eligible for open-label ZDV through this protocol. Modification of dose is recommended, however, patients who elect to continue current dose of ZDV after being informed of results of ACTG 019 will be allowed to do so. All patients enrolled in this study will continue to be followed until termination of this study. Above amendment added 11/01/89.

Study B: The wife or other female sexual partner is interviewed once at the beginning of the study and again when Study A is completed. The interview takes about 10 minutes and includes questions about the couple's sexual activity to help define the risk of becoming infected with HIV. In addition, blood is drawn to test for antibodies to HIV. The questionnaire and blood sample will be repeated at the time the patient is switched from blinded study therapy to open-label ZDV. (AMENDED 11/01/89) The results of the blood test are given to the person being tested. Information about the transmission of HIV and counseling are provided. It is recommended that the wife abstain from sexual contact with her husband, but if she does not, the use of condoms or condoms plus a spermicide is recommended. The decision about the type of precautions to take does not influence the opportunity to participate in the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed with caution for Study A:

* Hepatotoxic drugs.

Patients in Study A must have:

* Hemophilia with no symptoms for AIDS. Most patients will have well-established factor 8 or 9 deficiency. However, patients with other coagulation diseases, such as factor 5 deficiency, and von Willebrand disease, will also be acceptable for the study.

Wives in Study B are included even if they are known to be seropositive or are not sexually active at the time the study starts.

Prior Medication:

Allowed for Study A:

* Patients who were on the Phase I ZDV study, ACTG 017, or are on ACTG 062 may enter after waiting 3 weeks.

Exclusion Criteria

Co-existing Condition:

Patients in Study A with the following symptoms or conditions are excluded:

* AIDS-defining illness.
* Severe ARC.
* Severe or prolonged toxicity.

Concurrent Medication:

Excluded for Study A:

* Isoniazid or rifampin.
* Treatment for Pneumocystis carinii pneumonia (PCP), oral candidiasis, and localized cutaneous herpes simplex or zoster infections.
* Probenecid.
* Aspirin on a regular basis, or for more than 72 hours without contacting the investigator.
* Drugs causing neutropenia or significant risk of nephrotoxicity.

Patients in Study A with the following prior conditions are excluded:

* AIDS-defining opportunistic infection or malignancy.
* Unexplained temperature greater than 38 C for more than 5 consecutive days or more than 10 days in any 30-day period in the 2 years prior to entry.
* Unexplained diarrhea defined as three or more liquid stools per day, persisting more than 7 days within 2 years prior to entry.
* Unintentional weight loss of greater than 10 lbs. or more than 10 percent of usual body weight within 2 years prior to study entry.
* Oral hairy leukoplakia at any time prior to entry.
* Oral candidiasis unrelated to the use of antibiotic therapy for more than 2 weeks within 2 years prior to entry or within the past 3 months.
* Herpes zoster within 2 years prior to entry into the study.

Prior Medication:

Excluded for Study A:

* Antiretroviral agents, including ZDV, ribavirin, HPA-23, rifampin, AL721 within 8 weeks of study entry.
* Significant course of immunomodulating agents such as steroids (greater than 1 week), isoprinosine, thymic factors within 3 months of study entry.
* Any other experimental therapy within 3 months of study entry.

Discouraged but not forbidden for Study B:

* Sexual contact with infected husband.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 538
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Merigan, Study Chair
Locations (23):
- United States (23):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford Univ School of Medicine, Stanford, California
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Price W, Merigan T, Peterman T. Condom usage reported by female sexual partners of asymptomatic HIV seropositive hemophilic men. Int Conf AIDS. 1989 Jun 4-9;5:420 (abstract no ThBP30)